CLINICAL TRIAL: NCT03418974
Title: Safety and Efficacy of Statins for Chinese Patients With Dyslipidemia: A Network Register-based Follow-up Study
Brief Title: Safety and Efficacy of Statins for Chinese Patients With Dyslipidemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Collaborators: Peking University People's Hospital (Other); Jiangsu Wanbang Medicine Marketing Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Jinming Yu, Professor of School of Public Health, Fudan University, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BZ1701
Record Dates: First submitted 2018-01-14; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Dyslipidemias
Keywords: Dyslipidemia; Cardiovascular Diseases; Hypertension; LDL-C
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; Hypertension | interventions — pitavastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pitavastatin treatment (Experimental): The drug pitavastatin is given to the patient according to the doctor's order and restricted to BangZhi produced by Jiangsu Wanbang Medicine Marketing Co., Ltd..
  Interventions: Drug: Pitavastatin
- Atorvastatin treatment (Experimental): The drug atorvastatin is given to the patient according to the doctor's order and the drug band is unspecified.
  Interventions: Drug: Atorvastatin
- Rosuvastatin treatment (Experimental): The drug atorvastatin is given to the patient according to the doctor's order and the drug band is unspecified.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Pitavastatin — Capsule/Tablet, oral, follow the doctor's advice Participants will receive pitavastatin treatment for 3 or 12 weeks.
  Arms: Pitavastatin treatment
Drug: Atorvastatin — Capsule/Tablet, oral, follow the doctor's advice Participants will receive atorvastatin treatment for 3 or 12 weeks.
  Arms: Atorvastatin treatment
Drug: Rosuvastatin — Capsule/Tablet, oral, follow the doctor's advice Participants will receive rosuvastatin treatment for 3 or 12 weeks.
  Arms: Rosuvastatin treatment

SUMMARY:
This study is designed to verify the clinical efficacy and safety of different statins in dyslipidemia patients, and explore the effects on glycometabolic in patients with impaired glucose regulation.

DETAILED DESCRIPTION:
Study Objective:

1. The main Objective: To explore the effects of different statins lipid-lowering treatment on glucose metabolism in patients with impaired glucose regulation in a large sample of Chinese population;
2. The secondary Objective: To obtain real-world evidence of the clinical efficacy and safety of statins lipid-lowering therapy in Chinese patients.

Study Design: The study was an open-label, multi-center network register-based follow-up study.

The total sample size: 10000 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of ASCVD (Acute coronary syndrome, Stable coronary heart disease, Postoperative revascularization, Ischemic cardiomyopathy, Ischemic stroke, Transient ischemic attack, Peripheral atherosclerotic disease).
2. ASCVD overall risk assessment for high-risk groups: Diabetic patients with LDL-C≥1.8mmol/L（70mg/dl）and age was equal or greater than 40 years old;
3. Patients with hypertension, LDL-C > 2.6mmol/L (100mg/dL) and combined with at least two risk factors. Risk factors include smoking, low HDL-C (HDL-C<1mmol/L, 40mg/dL), male aged over 45 years old or female aged over 55 years old; *** The above (1)-(3) are juxtapositions, patients can be included into the group if only they are satisfied with at least one of the inclusion criteria.

Exclusion Criteria:

1. Patients with any allergy to statins;
2. ACS patients in acute stage；
3. Patients with severe liver disease or biliary obstruction；
4. Patients taking cyclosporine；
5. Patients who have being treated with statins currently or in the past;
6. Pregnant or lactating women and those women who planning to be pregnant;
7. Immunodeficiency or Immunocompromised patients;
8. Patients with hypothyroidism (expect those patients whose thyroid function returned to normal level after drug therapy);
9. Patients using systemic hormone drug;
10. Researchers decided that the patients who was not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
LDL-C target achieving rate | 3 months
  To measure the levels of LDL-C in mmol/L and calculate the LDL-C target achieving rate.

SECONDARY OUTCOMES:
Blood lipid parameters | 3 months
  The levels of total cholesterol (TC) in mmol/L
Blood lipid parameters | 3 months
  The levels of triglyceride (TG) in mmol/L
Blood lipid parameters | 3 months
  The levels of low density lipoprotein cholesterol (LDL-C) in mmol/L
Blood glucose levels | 1 year
  To measure the level of glycosylated hemoglobin (HbA1) in percent (%)
Fasting blood glucose | 1 year
  The levels of fasting blood glucose (FBG) in mmol/L
Blood lipid parameters | 1 year
  The levels of total cholesterol (TC) in mmol/L
Blood lipid parameters | 1 year
  The levels of triglyceride (TG) in mmol/L
Blood lipid parameters | 1 year
  The levels of low density lipoprotein cholesterol (LDL-C) in mmol/L
Blood lipid parameters | 1 year
  The levels of High density lipoprotein cholesterol (HDL-C) in mmol/L
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 1 year
  To evaluate the safety and tolerability of the three statins, the incidence of treatment-emergent adverse events should be recorded though the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Jin, Professor, Principal Investigator — School of Public Health，Fudan University; Dayi Hu, Professor, Principal Investigator — Director of Department of Cardiology, Peking University People's Hospital; Director of Institute of Cardiovascular Disease, Peking University
Locations (2):
- China (2):
  - Heart Center of Peking University People's Hospital, Beijing, Beijing Municipality
  - School of Public Health, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No